CLINICAL TRIAL: NCT01625949
Title: Study of Stem Cell Therapy in Patients With Myocardial Infarction and Persistent Total Occlusion of Infarct Related Artery
Brief Title: Stem Cell Therapy in Patients With Myocardial Infarction and Persistent Total Occlusion of Infarct Related Artery
Acronym: COAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Sandeep Seth, Additional Professor, Department of Cardiology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICMR project 80/3/2010-BMS; I-676 (Other Grant/Funding Number: Indian council of medical research)
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Acute Myocardial Infarction
Keywords: myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Standard Therapy) (Active Comparator): Control Arm Receiving The Standard Therapy including successful coronary intervention and stenting
  Interventions: Procedure: coronary dilatation and stenting
- Intracoronary stem cells (Experimental): Intracoronary stem cells will be injected in the infarct related artery after a successful coronary dilatation and stenting
  Interventions: Procedure: Intracoronary stem cells injection

INTERVENTIONS:
Procedure: Intracoronary stem cells injection — Intracoronary stem cells will be injected in the infarct related artery after a successful coronary dilatation and stenting autologous bone marrow stem cells from iliac crest 60 ml bone marrow will be extracted and purified for mononuclear cells which will be injected.
  Arms: Intracoronary stem cells
Procedure: coronary dilatation and stenting — coronary dilatation and stenting
  Arms: Control Arm (Standard Therapy)

SUMMARY:
Background: When an acute myocardial infarction occurs, the artery supplying the infarct zone should be opened within twenty four hours of onset of infarction. This has clearly been shown to be beneficial.

If the patient presents later than 24 hours of onset, at that stage a large part of the damage to the heart is irreversible. Intervening at this stage (beyond 24 hours is controversial). Some trials suggest that opening the artery even at this stage positively modifies the remodeling process while other trials suggest that such a benefit is not seen.

Hypothesis: Opening an infarct related artery after 24 hours (until 6 months) and combining it with intracoronary stem cell therapy may provide incremental benefit.It is possible that the lack of benefit seen with late revascularization (>24 hrs) after MI may be offset by giving intracoronary stem cells after opening the artery.

DETAILED DESCRIPTION:
Objectives

The benefit of opening an infarct related artery after the period of myocardial salvage (In patients who do not come to medical attention within 24 hrs of an infarctions) has been questioned in recent trials. On the other hand, Stem cell therapy after myocardial infarction has been shown to improve myocardial function both in the acute and chronic phases. It is possible that the lack of benefit seen with late revascularization (>24 hrs) after MI may be offset by giving intracoronary stem cells after opening the artery. Patients with recent myocardial infarction (MI) and occluded infarct related arteries supplying a large myocardial territory and with reduced ejection fraction will be randomized to a percutaneous coronary intervention (PCI) arm and a PCI plus stem cell arm .

The objective of the trial is to demonstrate that opening an infarct related artery after 24 hours and before six months and following it with intracoronary stem cell therapy may provide incremental benefit.

The primary objective

To demonstrate benefits in left ventricular recovery (improvement in function by echocardiogram and Nuclear imaging: Multigated acquisition [MUGA], reduction in scar size by tetrofosmin scan/Positron Emission Tomography[PET]. )

The secondary objectives

To demonstrate improvement in functional capacity as assessed by 6 minute walk test and quality of life assessment, along with reduction of first occurrence of recurrent MI, hospitalization/treatment of New York Heart Association class IV congestive heart failure, or death

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 80 years
2. Sex:Both
3. Recent MI (3-28 d)
4. Obstructed artery needing intervention
5. consent for stem cell therapy

Exclusion Criteria:

1. Left main disease or Triple vessel disease[TVD] needing surgery
2. Hypotension
3. Consent not given

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
left ventricular function | 3 Months
  Change in left ventricular function (assessed by Nuclear imaging and ECHO) and change in myocardial viability [assessed by PET].

SECONDARY OUTCOMES:
change in functional capacity | 3 months
  change in functional capacity as assessed by 6 minute walk test, quality of life assessment, first occurrence of recurrent MI,

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Seth, DM, Principal Investigator — All India Institute of Medical Sciences; Balram Airan, DM, Study Chair — All India Institute of Medical Sciences; V K Bahl, DM, Study Chair — AIIMS, New Delhi; Balram Bhargava, DM, Study Chair — AIIMS, New Delhi; Chetan Patel, Study Chair — AIIMS, New Delhi; Sujata Mohanty, Study Chair — AIIMS, New Delhi; Rajiv Narang, DM, Study Chair — AIIMS, New Delhi; S Ramakrishnan, DM, Study Chair — AIIMS, New Delhi; K C Goswami, DM, Study Chair — AIIMS, New Delhi; Rakesh Yadav, DM, Study Chair — AIIMS, New Delhi; Ambuj Roy, DM, Study Chair — AIIMS, New Delhi; G Karthikeyan, DM, Study Chair — AIIMS, New Delhi; Gautam Sharma, DM, Study Chair — AIIMS, New Delhi; Sandeep Singh, DM, Study Chair — AIIMS, New Delhi; Sandeep Mishra, DM, Study Chair — AIIMS, New Delhi; Nitish Naik, DM, Study Chair — AIIMS, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, India

REFERENCES:
- [Background] Strauer BE, Brehm M, Zeus T, Bartsch T, Schannwell C, Antke C, Sorg RV, Kogler G, Wernet P, Muller HW, Kostering M. Regeneration of human infarcted heart muscle by intracoronary autologous bone marrow cell transplantation in chronic coronary artery disease: the IACT Study. J Am Coll Cardiol. 2005 Nov 1;46(9):1651-8. doi: 10.1016/j.jacc.2005.01.069. PMID 16256864
- [Background] Menasche P, Alfieri O, Janssens S, McKenna W, Reichenspurner H, Trinquart L, Vilquin JT, Marolleau JP, Seymour B, Larghero J, Lake S, Chatellier G, Solomon S, Desnos M, Hagege AA. The Myoblast Autologous Grafting in Ischemic Cardiomyopathy (MAGIC) trial: first randomized placebo-controlled study of myoblast transplantation. Circulation. 2008 Mar 4;117(9):1189-200. doi: 10.1161/CIRCULATIONAHA.107.734103. Epub 2008 Feb 19. PMID 18285565
- [Background] Dib N, Michler RE, Pagani FD, Wright S, Kereiakes DJ, Lengerich R, Binkley P, Buchele D, Anand I, Swingen C, Di Carli MF, Thomas JD, Jaber WA, Opie SR, Campbell A, McCarthy P, Yeager M, Dilsizian V, Griffith BP, Korn R, Kreuger SK, Ghazoul M, MacLellan WR, Fonarow G, Eisen HJ, Dinsmore J, Diethrich E. Safety and feasibility of autologous myoblast transplantation in patients with ischemic cardiomyopathy: four-year follow-up. Circulation. 2005 Sep 20;112(12):1748-55. doi: 10.1161/CIRCULATIONAHA.105.547810. PMID 16172284
- [Background] Assmus B, Fischer-Rasokat U, Honold J, Seeger FH, Fichtlscherer S, Tonn T, Seifried E, Schachinger V, Dimmeler S, Zeiher AM; TOPCARE-CHD Registry. Transcoronary transplantation of functionally competent BMCs is associated with a decrease in natriuretic peptide serum levels and improved survival of patients with chronic postinfarction heart failure: results of the TOPCARE-CHD Registry. Circ Res. 2007 Apr 27;100(8):1234-41. doi: 10.1161/01.RES.0000264508.47717.6b. Epub 2007 Mar 22. PMID 17379833